CLINICAL TRIAL: NCT03929042
Title: Evaluating the Effectiveness of Posture Correction Girdle for Adolescents With Early Scoliosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr. Kenny Kwan, Clinical Assistant Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW16-505
Record Dates: First submitted 2017-07-18; First posted 2019-04-26 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: AIS

STUDY DESIGN:
Intervention Model Description: Patients currently on underarm brace treatment will be eligible for participation in our study. For those that agree to participate, a AP/lat standing X-ray and force measurements of the brace on the rib and loin hump will be taken. They will be then be asked to wear a customised postural correction girdle 24 hours after they have taken off the brace. The same study assessments will be conducted.
  Patients whose forces and radiological Cobb correction are comparable between the two methods of treatment will be given a choice to either continue the hard brace or wear the posture correction girdle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Posture Correction Girdle (Experimental): Our research team has designed a prototype of posture correction girdle based on the clinical, textile science, material and ergonomics engineering analyses as an alternative to hard brace for AIS. The design of the posture correction girdle incorporates different mechanisms, such as 1) compression and pulling forces through a close fit of the intimate apparel, 2) lumbar flexion by using supporting belt, 3) transverse forces applied by inserting pads inside the pocket lining by using the principle of the 3-point pressure system.
  Interventions: Device: Posture correction girdle

INTERVENTIONS:
Device: Posture correction girdle — Our research team has designed a prototype of posture correction girdle based on the clinical, textile science, material and ergonomics engineering analyses as an alternative to hard brace for AIS. The design of the posture correction girdle incorporates different mechanisms, such as 1) compression and pulling forces through a close fit of the intimate apparel, 2) lumbar flexion by using supporting belt, 3) transverse forces applied by inserting pads inside the pocket lining by using the principle of the 3-point pressure system.

SUMMARY:
Through the ITF-Tier 3 project (ITS/ 237/ 11), a prototype of the posture correction girdle based on the clinical, textile science, material and ergonomics engineering analyses has been developed for preteen and teenage girls aged 10 to 13 who have the early stages of scoliosis. The girdle provides a corrective force onto the torso by the warping and elastic extension of the shoulder straps and waistband and the insertion of semi-rigid EVA padding and uses a point-pressure support system to achieve the target of posture improvement and spinal progression control with physical and psychological comfort.

In order to evaluate the effectiveness of the posture correction girdle, it is proposed to recruit 10 patients to take low dose x-ray (sterEOS) at QMH at supine position. Then, the patient should wear the girdle for two hours and take another x-ray at standing position. If the Cobb's angle of the patient on girdle at standing position can be same as her supine position. It can prove the effectiveness of the girdle.

DETAILED DESCRIPTION:
Background Information Scoliosis in patients between 10 and 18 years of age is termed adolescent scoliosis. The most common type of scoliosis is one of which the cause is not known. This is called "idiopathic" or "adolescent idiopathic scoliosis (AIS)". The main risk factors of curve progression could be skeletal immaturity, female gender and large curve magnitude. It has been found that nearly 10% of all adolescents have some degree of spinal curve or deformity after their tenth year. The health of patients, such as cardiac and pulmonary functions, may be affected if their spinal deformity is very serious. Hence, the most ideal way is to monitor and control spinal curvature once AIS has been found.

Treatment options for scoliosis In general, patients are suggested to undergo different types of treatments according to their spine situations and stage of scoliosis. Surgery is suggested for patients with spinal curves that are greater than 41-50 degrees, while bracing is a non-invasive treatment suggested for those with spinal curves between 21-40 degrees. Thoraco-lumber-sacral-orthosis (TLSO) or cervico-thoraco-lumbo-sacral orthosis (CTLSO) braces are the most commonly prescribed and used braces. The 3-point pressure system is primarily applied by all TLSO braces in order to correct the spinal curve and reduce the curve progression. The plaster cast is tailor-made according to the body shape of each patient. The upper torso of the wearer needs to be tightly compressed by this non-breathable material for 23 hours every day. The duration of the treatment duration will be for years until the bones are fully mature.

Aside from the fact that newer types of flexible brace products in the market are not available in large numbers, their effectiveness continues to be controversial and there is much room for improvement. The SpineCor Dynamic brace is one of the flexible braces used to treat AIS. The theory behind the SpineCor system is known as spinal coupling. Spinal coupling corrects deformities by reversing abnormal posture and body shape into their opposite position so that the abnormal alignment of the spine can be corrected. As the spinal curve of each patient is different, thus appropriate positions and tensions of the elastics will be respectively placed and adjusted by a professional before the patient wears the brace. It has been found that the curve progression rate of those who wear the SpineCor Dynamic brace is significantly higher than those who wear the rigid brace. It is believed that the ineffectiveness of the flexible brace may be caused by the shifting of the elastic bands. The elastic bands present on the brace are not fixed to the body of the wearer, and may easily shift to other areas during movement. Hence, the corrective force will no longer be exerted onto the correct position for posture and body shape correction.

A summary of the research rationale is listed below. Research rationale 1: Low treatment compliance Treatment through the use of a hard brace has low compliance due to discomfort and psychological issues, such as an awkward and bulky appearance. Flexible braces have other issues, such as discomfort caused by the elastic bands, inconvenience when going to the toilet, and unusual designs, which also result in low compliance. New designs that aim to improve compliance are therefore extremely important.

Research rationale 2: Limited product choice for adolescents with early scoliosis Hard brace treatment is overly excessive for adolescents with early scoliosis due to the high corrective force which nearly constrains all movements. The flexible brace treatment is an alternative option; however, its efficacy remains controversial. Intimate apparel that has a specialized design for teenagers with scoliosis is limited and a large majority can only provide some improvement for poor postures, such as hunchback. A scientific approach should be used to design and develop functional intimate apparel as a treatment option for adolescents with early scoliosis.

ELIGIBILITY:
Inclusion Criteria:

* • Satisfy SRS criteria for bracing15

  * Curretly treated for rigid underarm brace
  * Primary Cobb angle between 25 to 40 degrees

Exclusion Criteria:

* • Contraindications for x-ray exposure

  * Diagnosis of other musculoskeletal or developmental illness that might be responsible for the spinal curvature
  * History of previous surgical or orthotic treatment for AIS
  * Contraindications for pulmonary and / or exercise tests
  * Psychiatric disorders
  * Recent trauma
  * Recent traumatic (emotional) event

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2017-07-17 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Measure the spinal correction of posture correction girdle and hard brace | 2 weeks
  The Cobb angle (unit: degree) of posture correction girdle and hard brace will be compared and reported.

SECONDARY OUTCOMES:
Measure the pressure forces exerted by posture correction girdle and hard brace | 2 weeks
  The pressure forces (unit: kpa) of posture correction girdle and hard brace will be compared and reported.
Measure the spinal correction of posture correction girdle after 6 months | 6 months
  The Cobb angle (unit: degree) after 6-month of posture correction girdle treatment will be calculated and reported.
Measure the pressure changes of posture correction girdle after 6 months | 6 months
  The pressure forces (unit: kpa) after 6-month of posture correction girdle treatment will be calculated and reported.
Measurement of patient-related outcome of posture correction girdle and hard brace by EQ-5D-5L | 6 months
  Health-related quality of life, Euroqol (EQ-5D-5L)
  The descriptive system comprises 5 dimensions in 5 questions. Each dimension has 5 levels which ranges from 0-no problems to 4-extreme problems. Total score is ranged from 0 to 20. The higher values represent a worse outcome.
Measurement of patient-related outcome of posture correction girdle and hard brace by SRS-22 | 6 months
  Health-related quality of life (SRS-22)
  The questionnaire consists of 22 questions and each question has 5 levels. The maximum score in each domain is 5 (greatest quality) and minimum score is 1 (poorest quality). Total score is ranged from 22 to 110. The higher values represent a better outcome.
Measurement of patient-related outcome of posture correction girdle and hard brace by TAPS | 6 months
  Patients' perception of self-image (TAPS)
  The TAPS included 3 sets of figures that depict the trunk from 3 viewpoints. Drawings are scored from 1 (greatest deformity) to 5 (smallest deformity). A mean score ranged from 1 to 5 is obtained. The higher mean scores represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Kenneth Cheung, MBBS (UK), MD (HK), Study Chair — The University of Hong Kong
Locations (1):
- Duchess of Kent Children's Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No